CLINICAL TRIAL: NCT05700656
Title: Phase I/II Study With Galunisertib Combined With Capecitabine in Patients With Advanced Chemotherapy Resistant Colorectal Cancer With Peritoneal Metastases
Brief Title: Galunisertib Combined With Capecitabine in Advanced CRC With PM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Amsterdam UMC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M22TGA
Record Dates: First submitted 2023-01-03; First posted 2023-01-26 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer Metastatic; Peritoneal Carcinomatosis
Keywords: colorectal cancer; metastatic colorectal cancer; peritonitis carcinomatosa
MeSH Terms: conditions — Peritoneal Neoplasms; Colorectal Neoplasms | interventions — LY-2157299; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Galunisertib plus capecitabine (Experimental): Galunisertib 150 mg BID for 14 days in a 28-day cycle plus capecitabine 1000 mg/m2 BID for 14 days in a 28-day cycle
  Interventions: Drug: Galunisertib plus capecitabine

INTERVENTIONS:
Drug: Galunisertib plus capecitabine — Combination therapy with galunisertib plus capecitabine

SUMMARY:
This is a two-center open-label non-randomized proof of principle study consisting of a dose-finding part (phase I) and phase II study with Simon two-stage design investigating the anti-tumor activity of the combination of capecitabine and galunisertib in patients with colorectal cancer with peritoneal metastases.

DETAILED DESCRIPTION:
This is a two-center pharmacological open-label non-randomized proof of principle study consisting of two parts: a phase I study evaluating the RP2D of galunisertib in combination with capecitabine; and a phase II study investigating the anti-tumor activity and safety of galunisertib in combination with capecitabine in advanced colorectal cancer (CRC) with peritoneal metastases (PM).

In phase II of the study a Simon two-stage design will be used. 15 patients will be treated with the galunisertib/capecitabine combination. If at least 2 out of 15 patients respond, an additional cohort of 10 patients will be included to a total of 25 patients. With 6 or more responses, the treatment will be declared to be of sufficient activity and with 5 or less it will be declared of insufficient activity.

The galunisertib dose will be 150 mg twice daily (BID) for the first 14 days of every 4-week cycle, which is the maximum tolerated dose when given as single agent (except of day 1 of cycle 1: single dose of galunisertib 150 mg for PK analysis, from day 2: 150 mg BID).

Capecitabine will be dosed during every 14-day on time of galunisertib at 1000 mg/m2 BID, which is the labelled dose as monotherapy and will in case of toxicities be reduced according to standard care.

Clinical assessments will be performed routinely to monitor safety. Anti-tumor activity will be measured by CT scan according to RECIST 1.1 criteria. Tumor biopsies will be obtained for exploratory objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological proof of CRC with at least confirmed peritoneal metastases (presence of additional extraperitoneal metastases is allowed);
2. Disease progression or relapse upon treatment for advanced CRC with fluoropyrimidine containing chemotherapy as single agent or in combination with other anti-cancer drugs, with no treatment options at time of inclusion (combinations with oxaliplatin, irinotecan, bevacizumab and cetuximab/panitumumab are allowed);
3. Age ≥ 18 years;
4. Able and willing to give written informed consent and informed consent form must have been signed before start of the trial;
5. WHO performance status of ≤1;
6. Able and willing to undergo blood sampling for PK analysis;
7. Able and willing to undergo tumor biopsy before start, during treatment and at the end of treatment;
8. Life expectancy > 3 months allowing adequate follow up of toxicity and anti-tumor activity;
9. Evaluable disease according to RECIST 1.1 criteria (measurable disease for the phase II part; evaluable disease is sufficient for the phase I part);
10. Minimal acceptable safety laboratory values

    1. ANC of ≥1.5 x 109/L
    2. Platelet count of ≥100 x 109/L
    3. Hepatic function as defined by serum bilirubin ≤ 1.5 x ULN, ALAT and ASAT ≤ 3.0 x ULN, or ALAT and ASAT < 5 x ULN in patients with liver metastases
    4. Renal function as defined by serum creatinine ≤ 1.5 x ULN
    5. Creatinine clearance ≥ 50 ml/min (by Cockcroft-Gault formula or MDRD);
11. Negative pregnancy test (urine or serum) for female patients with childbearing potential.
12. Able and willing to swallow tablets.

Exclusion Criteria:

1. Any treatment with investigational drugs within 30 days prior to receiving the first dose of investigational treatment and/or radio- or chemotherapy within the last 2 weeks prior to receiving the first dose of investigational treatment. Palliative radiation (1x 8Gy) is allowed; except radiotherapy focused on the liver;
2. Known or suspected complete or partial dihydropyrimidine dehydrogenase deficiency (Mutant for DPD*2A genotype, 1236G>A genotype, 1679T>G genotype and 2846A>T genotype);
3. Symptomatic or untreated leptomeningeal disease;
4. Symptomatic brain metastasis. Patients previously treated or untreated for these conditions that are asymptomatic in the absence of corticosteroid therapy are allowed to enrol. Brain metastasis must be stable with verification by imaging (e.g.

   brain MRI or CT completed at screening demonstrating no current evidence of progressive brain metastases). Patients are not permitted to receive enzyme inducing anti-epileptic drugs or corticosteroids;
5. History of cardiac disease, including myocardial infarction within 6 months before first dose of study medication, unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, or uncontrolled hypertension, major cardiac abnormalities, a predisposition for developing aneurysms including family history of aneurysms, Marfan syndrome, bicuspid aortic valve, or evidence of damage to the large vessels of the heart;
6. Treatment with CYP3A4 inducers or inhibitors and/or concomitant treatment with CYP2C9 substrates with narrow therapeutic window, including but not limited to vitamin K antagonizing anticoagulants (e.g. acenocoumarol, phenprocoumon and warfarin) and phenytoin is not allowed;
7. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral galunisertib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, major small bowel surgery);
8. Woman who are pregnant or breast feeding;
9. Patients who have undergone any major surgery within the last 2 weeks prior to starting study drug or who would not have fully recovered from previous surgery;
10. Active infection requiring systemic antibiotics or uncontrolled infectious disease;
11. Patients with a known history of hepatitis B or C or known Human Immunodeficiency Virus HIV-1 or HIV-2 type patients;
12. Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for the study;
13. Known hypersensitivity to one of the study drugs or excipients.
14. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of <1% per year (when used consistently and correctly) during the treatment period and for at least 90 days after the last dose of galunisertib and/or capecitabine.
15. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events according to CTCAE v5.0, dose limiting toxicities | 28 days
  To determine the safety and RP2D of galunisertib plus capecitabine in patients with advanced chemotherapy resistant CRC with peritoneal metastases
Objective response rate (ORR) | through study completion, an average of 6 months per patient
  To determine the anti-tumor activity as measured by ORR of galunisertib plus capecitabine in patients with advanced chemotherapy resistant CRC with PM.

SECONDARY OUTCOMES:
Duration of response (DOR) | through study completion, an average of 6 months per patient
  Time from first response until progression
Time to response (TTR) | From date of study entry until first objective response, an average of 2 months
  Time from start of treatment until first objective response
Progression free survival (PFS) | From date of study entry until the date of first documented progression of date of death from any cause, whichever comes first, assessed up to 5 years
  Time from start of the treatment until progression
Overall survival (OS) | From date of study entry until date of death from any cause, assessed up to 5 years
  Time from start of the study until death
Cmax, Tmax, AUC, T0.5, MTD | 14 days
  Pharmacokinetic profile of galunisertib
RNA sequencing, THG-b signaling, other | through study completion, an average of 2 years
  Exploratory genomic analyses to determine biomarkers for response and resistance to the combination of galunisertib and capecitabine

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - Amsterdam UMC, Amsterdam

IPD SHARING:
Plan to Share IPD: Undecided